CLINICAL TRIAL: NCT06290362
Title: The New Age of Cyber Care: Exploring Digitalized Interventions for Stress and Problem Solving - A Randomized Controlled Trial
Brief Title: Exploring Digitalized Interventions for Stress and Problem Solving
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gizem Beycan Ekitli, PhD., Research Assistant Dr., Ege University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: EgeTrial4
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Stress; Problem-solving
Keywords: telemedicine; internet-based intervention; stress; problem-solving

STUDY DESIGN:
Intervention Model Description: The current 8-week randomized, single-blind factorial trial was conducted with a control group and one intervention group. Over eight weeks, participants received cognitive behavioral-based intervention through online sessions. Pre-/post-test and follow-up assessments employed.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Any intervention applied. Following the completion of the research, the need for psychosocial support among the control group participants was assessed, and it was found that none of the students in the control group required such support.
- Cognitive Behavioural Theory-based group consultation (Experimental): Cognitive Behavioural Theory-based group consultation was given to the intervention group through an Instagram as online social media platform. This approach has been developed with the philosophy of Cognitive Behavioral Theory (Eskin, 2009). For three days a week over eight weeks of intervention conducted with synchronized psychoeducation sessions, online posts, surveys, personal sharing messages, and group interaction tools.
  1. Introduction and warm-up,
  2. Problem orientation-identifying the problem,
  3. Identifying prior problems-Which one I want to start?
  4. Recognizing the losses caused by problems and complaints,
  5. Setting reachable and realistic goals,
  6. Generating alternatives-What can I do?
  7. Regulating emotions,
  8. Experimenting and exploring. Sessions were completed in approximately one hour as semi-structured interactive group training according to group dynamics.
  Interventions: Behavioral: Cognitive Behavioural Theory-based group consultation

INTERVENTIONS:
Behavioral: Cognitive Behavioural Theory-based group consultation — Cognitive Behavioural Theory-based group consultation was given to the intervention group through an Instagram as online social media platform. This approach has been developed with the philosophy of Cognitive Behavioral Theory (Eskin, 2009).
  For three days a week over eight weeks, informative posts were shared, asynchronous testing and self-discovery activities were carried out, and a synchronous tele-psychoeducation session was held once a week. The participants were connected to the live broadcast of the research team, and they interacted via text messages. In this interaction, further suggestions related to the goals of the week were given, previous assignments were checked, homework for the next session was given, personal experiences and the needs of the participants were determined, and necessary feedback was provided. Instagram had the feature of maintaining the records of all participants' attendance at these events.
  Arms: Cognitive Behavioural Theory-based group consultation

SUMMARY:
Excessive and prolonged stress can have detrimental effects on both psychological and physiological health, compromising overall well-being and functioning. This study examines the impact of telepsychiatric group consultation using Instagram as an unexplored online social media platform on stress levels and problem-solving skills among young adults.

DETAILED DESCRIPTION:
A randomized, single-blind factorial trial with a control group was conducted. Over eight weeks, participants received cognitive behavioral-based intervention through online sessions. Pre-/post-test and follow-up assessments employed the Problem-Solving Inventory and Perceived Stress Scale, analyzed using factorial analysis of variance. Effect sizes were determined using ηp2 and Cohen's r.

Significant differences were found between groups for Problem-Solving Inventory (F(2-104):5.005)(p<0.05). The key findings of our RCT study is the strong impact of digitalized intervention on the time-group interaction (p<0.05). This highlights the effectiveness of the Instagram-based telehealth tool in facilitating long-lasting improvements among young adults. These findings shed light on the potential of social media platforms, like Instagram, as not only popular but successful tools for mental health interventions. Nurses can incorporate these digital interventions to enhance mental health support, reach a wider audience, and overcome barriers associated with traditional methods.

1. H1: There is a significant difference between the mean scores of the Problem Solving Inventory in favour of the Instagram-based intervention group in the time series.
2. H1: There is a significant difference between the mean scores of the Perceived Stress Scale in favour of the Instagram-based intervention group in the time series.
3. H1: Instagram-based telehealth is effective for reducing Problem Solving Inventory scores.
4. H1: Instagram-based telehealth is effective for reducing Perceived Stress Scale scores.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age,
* Being an university student,
* Volunteer for the study,
* Possess the necessary technological resources

Exclusion Criteria:

* Have a physical or sensory impairment that would affect the ability to use online technology (e.g., history of temporal brain damage, limb loss, hearing loss, etc.),
* Have a psychiatric diagnosis that would affect decision-making and orientation assessment abilities
* Be receiving any professional support that could potentially influence their coping skills during data collection

This calculation was performed to ensure that the study would have an appropriate sample size to detect meaningful effects and draw reliable conclusions. In this study, an alpha level of 0.05 and a beta level of 0.20 have been set. Based on the results of previous similar studies, it has been determined that a minimum sample size of 24 (total 48) is required for each group.

Following the completion of the announcement and registration phase, a random assignment process was conducted to allocate 54 students into either the control or intervention groups, adhering to the guidelines of the Consort Model.

Gender, problem-solving skills, and perceived stress levels were taken into account during the group allocation process.

The RCT's statistical power, calculated post hoc within a 95% confidence interval and a sampling error of d=.05, was determined to be 83.0%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (first evaluation with posttest) | Through intervention completion, an average of 2 month
  The Perceived Stress Scale is designed to measure how stressful situations in one's life are perceived. The five-point Likert-type scale items (0-never, 4-very often) are interpreted over the total score and two sub-dimensions (insufficient self-efficacy and stress disturbance perception). A high total score indicates that the person perceives the stress he/she has been loaded with as high; it is interpreted as the methods used in coping with stress are not functional, and therefore they cannot cope with stress effectively. In our study, the Cronbach's alpha coefficient of the scale was determined as .75.
Problem Solving Inventory (first evaluation with posttest) | Through intervention completion, an average of 2 months
  The Problem Solving Inventory is a Likert-type scale, scored between 1 and 6, consisting of 35 items that measure adults' self-perception of problem-solving skills. There are items that are reverse coded and excluded from scoring. The scale's Turkish adaptation study's Cronbach alpha consistency coefficient was found to be .88. In our study, the Cronbach alpha coefficient was .78.The higher total scores obtained from the scale indicate that the individual perceives himself/herself as inadequate in terms of problem-solving skills.
Perceived Stress Scale (second evaluation with follow up) | Through intervention completion, an average of 5 month
  The Perceived Stress Scale is designed to measure how stressful situations in one's life are perceived. The five-point Likert-type scale items (0-never, 4-very often) are interpreted over the total score and two sub-dimensions (insufficient self-efficacy and stress disturbance perception). A high total score indicates that the person perceives the stress he/she has been loaded with as high; it is interpreted as the methods used in coping with stress are not functional, and therefore they cannot cope with stress effectively. In our study, the Cronbach's alpha coefficient of the scale was determined as .75.
Problem Solving Inventory (second evaluation with follow up) | Through intervention completion, an average of 5 months
  The Problem Solving Inventory is a Likert-type scale, scored between 1 and 6, consisting of 35 items that measure adults' self-perception of problem-solving skills. There are items that are reverse coded and excluded from scoring. The scale's Turkish adaptation study's Cronbach alpha consistency coefficient was found to be .88. In our study, the Cronbach alpha coefficient was .78.The higher total scores obtained from the scale indicate that the individual perceives himself/herself as inadequate in terms of problem-solving skills.

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Public data sharing is available for this study.
  beycan ekitli, gizem (2022), "Digitalization in Psychoeducation' The Effect of Tele-Psychoeducation", Mendeley Data, V1, doi: 10.17632/5g9bcjv43b.1
  http://dx.doi.org/10.17632/5g9bcjv43b.1
Supporting Information: Study Protocol, Analytic Code
Time Frame: By publication with no end date.
Access Criteria: It is planned to publish the research results in a high-impact journal in the field.
URL: http://dx.doi.org/10.17632/5g9bcjv43b.1